CLINICAL TRIAL: NCT05415488
Title: Dietary Treatment for IBS Within Primary Health Care
Acronym: KIPIBS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sahlgrenska University Hospital (Other)
Responsible Party: Principal Investigator, Magnus Simrén, Professor, Sahlgrenska University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022-01624-01
Record Dates: First submitted 2022-06-07; First posted 2022-06-13 (Actual); Last update posted 2023-12-01 (Actual); Status verified 2023-11

CONDITIONS: Irritable Bowel Syndrome
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Intervention Model Description: Intervention study with 2 parallel arms (1:1)
Who Masked: Participant
Masking Description: Participants will only be told that the both diets aim to relieve symptoms of IBS, and that none of the diets are expected to cure the disorder. No specific names of the diets will be given.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IBS dietary advice according to the NICE guidelines (Active Comparator): The traditional dietary advice according to the NICE guidelines and the systematic reviews performed by the British dietetic association (BDA) include having regular meals and to take time to eat, not to skip meals or eat too much at ones. The diet also limits intake of known trigger foods, such as coffee, alcohol, fizzy drinks, spicy foods, fatty foods etc. People who experience loose stools are recommended to avoid sweeteners (-ol), and people with wind/bloating are recommended to eat soluble fibers such as oats and flaxseeds.
  Interventions: Other: Online dietary group treatment
- A healthy diet according to the Swedish dietary guidelines (Sham Comparator): This diet includes eating 500 grams of vegetables and fruits/day, fish approximately 3 times/week, 70 grams of wholegrain/day and to limit intake of red meat.
  Interventions: Other: Online dietary group treatment

INTERVENTIONS:
Other: Online dietary group treatment — Dietary advice will be given during one 90 minute online group session

SUMMARY:
Irritable bowel syndrome (IBS) is a multifaceted disorder where diet plays a pivotal role in symptom generation and management. The traditional dietary advice given to patients in clinical settings are based on the NICE guidelines. Some of the advice included in these guidelines have limited scientific evidence. The aim of this study is to investigate the effectiveness of the traditional dietary advice in IBS, according to the NICE guidelines, within a primary health care setting, where treatment is delivered digitally and in groups of 8-12 individuals. As a sham comparator, one group will receive dietary advice according to the Swedish dietary guidelines regarding healthy eating habits.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with IBS (ROME IV) by physician
* Age 18-50
* Ability to read and understand Swedish
* Signed informed consent

Exclusion Criteria:

* Received dietary treatment for IBS previously
* Manifestations of other conditions that may explain gastrointestinal symptoms

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 240 (Estimated)
Dates: Start 2022-08-15 (Actual); Primary Completion 2024-09-15 (Estimated); Study Completion 2025-09-15 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with significant symptom reduction | From baseline vs. 6 weeks after group session
  A responder to treatment is defined as having a symptom reduction >50 measured by IBS-SSS

CONTACTS AND LOCATIONS:
Locations (1):
- Dept of Internal Medicine, Sahlgrenska University Hospital, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: Undecided